CLINICAL TRIAL: NCT06624293
Title: Access BNP Assay Clinical Subject Sample Collection Enrollment Study Protocol
Brief Title: Access BNP Clinical Enrollment Study
Status: Completed | Type: Observational
Sponsor: Beckman Coulter, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: BNP-05-24
Record Dates: First submitted 2024-09-18; First posted 2024-10-02 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-04

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — EDTA plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Subjects with heart failure: Targeting subjects in the acute care setting that present with suspicion of either new onset or worsening symptoms of heart failure
  Interventions: Diagnostic Test: BNP

INTERVENTIONS:
Diagnostic Test: BNP — Blood collected during this study will be tested on separate IUO BNP assay on a separate protocol. No active interventions will occur during this study.

SUMMARY:
The goal of this study is to collect blood from subjects with a suspicion of either new onset or worsened heart failure to be used for testing studies for a new product to aid in the diagnosis of heart failure.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide informed consent
* Adult greater than or equal to 22 years old, any gender, race, ethnicity
* Presenting with clinical suspicion of new onset heart failure or worsening symptoms suggestive of decompensated or exacerbated heart failure
* Ability to fulfill study data collection requirements (including responding to questions for the NYHA evaluation)

Exclusion Criteria:

* Individuals less than 22 years old
* Impairment in individual's capacity to give informed consent
* Dyspnea clearly not secondary to heart failure (e.g., primary lung disease or chest trauma).
* On dialysis
* On nesiritide infusion
* Subject clinical/medical history access is not available to Sponsor, delegates, and FDA or other regulatory agencies upon request.
* Active participation in a clinical study that may interfere with participation in this study (e.g., investigational drug study)
* Reason(s) determined by the Principal Investigator that would place the individual at increased risk or preclude the individual from fully complying with or completing the study.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study is expected to enroll approximately 1,100 subjects from intended use population. The study population (enrolled by the collective clinical sites) should reasonably represent the U.S. demographic population. Sponsor will monitor for age, race, gender representation A minimum of 400 subjects with a HF positive clinical site diagnosis need to be enrolled without being withdrawn/discontinued. Of the HF positive group, the sample size for severity assessment (> 80% power) requires a minimum of 340 subjects with a minimum of 50, 150, and 140 NYHA class II, III, and IV subjects, respectively, to detect a correlation between BNP level increase and the severity of heart failure.
Sampling Method: Non-Probability Sample
Enrollment: 1100 (Actual)
Dates: Start 2024-08-30 (Actual); Primary Completion 2025-02-18 (Actual); Study Completion 2025-02-18 (Actual)

PRIMARY OUTCOMES:
Heart failure positive subjects | During initial assessment in emergency department
  Subjects with BNP value above clinical decision point

SECONDARY OUTCOMES:
Heart failure negative subjects | During initial assessment in emergency department
  Subjects with BNP value below clinical decision point

CONTACTS AND LOCATIONS:
Locations (17):
- United States (17):
  - Loma Linda University Medical Center Department of Emergency Medicine, Loma Linda, California
  - UC Davis Health Department of Emergency Medicine, Sacramento, California
  - University of Florida College of Medicine, Gainesville, Florida
  - University of Florida College of Medicine - Jacksonville, Jacksonville, Florida
  - Indiana University Health, Indianapolis, Indiana
  - University of Kansas Medical Center Department of Emergency Medicine, Kansas City, Kansas
  - University of Maryland Baltimore University of Maryland Medical Center, Baltimore, Maryland
  - Henry Ford Health, Detroit, Michigan
  - Hcmc-Hhri, Minneapolis, Minnesota
  - University of New Mexico Department of Emergency Medicine, Albuquerque, New Mexico
  - Department of Emergency Medicine University of Rochester Medical Center, Rochester, New York
  - Department of Emergency Medicine Stony Brook University Medical Center, Stony Brook, New York
  - The Ohio State College of Medicine Department of Emergency Medicine, Columbus, Ohio
  - Medical University of South Carolina, Charleston, South Carolina
  - Vanderbilt University School of Medicine Center for Emergency Care Research and Innovation, Nashville, Tennessee
  - Ben Taub Hospital, Houston, Texas
  - University of Wisconsin Health University Hospital, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Long B, Koyfman A, Gottlieb M. Diagnosis of Acute Heart Failure in the Emergency Department: An Evidence-Based Review. West J Emerg Med. 2019 Oct 24;20(6):875-884. doi: 10.5811/westjem.2019.9.43732. PMID 31738714
- [Background] Fleg JL, Pina IL, Balady GJ, Chaitman BR, Fletcher B, Lavie C, Limacher MC, Stein RA, Williams M, Bazzarre T. Assessment of functional capacity in clinical and research applications: An advisory from the Committee on Exercise, Rehabilitation, and Prevention, Council on Clinical Cardiology, American Heart Association. Circulation. 2000 Sep 26;102(13):1591-7. doi: 10.1161/01.cir.102.13.1591. No abstract available. PMID 11004153
- [Background] Heidenreich PA, Bozkurt B, Aguilar D, Allen LA, Byun JJ, Colvin MM, Deswal A, Drazner MH, Dunlay SM, Evers LR, Fang JC, Fedson SE, Fonarow GC, Hayek SS, Hernandez AF, Khazanie P, Kittleson MM, Lee CS, Link MS, Milano CA, Nnacheta LC, Sandhu AT, Stevenson LW, Vardeny O, Vest AR, Yancy CW. 2022 AHA/ACC/HFSA Guideline for the Management of Heart Failure: A Report of the American College of Cardiology/American Heart Association Joint Committee on Clinical Practice Guidelines. J Am Coll Cardiol. 2022 May 3;79(17):e263-e421. doi: 10.1016/j.jacc.2021.12.012. Epub 2022 Apr 1. PMID 35379503
- [Background] Apple FS, Panteghini M, Ravkilde J, Mair J, Wu AH, Tate J, Pagani F, Christenson RH, Jaffe AS; Committee on Standardization of Markers of Cardiac Damage of the IFCC. Quality specifications for B-type natriuretic peptide assays. Clin Chem. 2005 Mar;51(3):486-93. doi: 10.1373/clinchem.2004.044594. PMID 15738513
- [Background] Maisel AS, Krishnaswamy P, Nowak RM, McCord J, Hollander JE, Duc P, Omland T, Storrow AB, Abraham WT, Wu AH, Clopton P, Steg PG, Westheim A, Knudsen CW, Perez A, Kazanegra R, Herrmann HC, McCullough PA; Breathing Not Properly Multinational Study Investigators. Rapid measurement of B-type natriuretic peptide in the emergency diagnosis of heart failure. N Engl J Med. 2002 Jul 18;347(3):161-7. doi: 10.1056/NEJMoa020233. PMID 12124404
- [Background] Ponikowski P, Voors AA, Anker SD, Bueno H, Cleland JG, Coats AJ, Falk V, Gonzalez-Juanatey JR, Harjola VP, Jankowska EA, Jessup M, Linde C, Nihoyannopoulos P, Parissis JT, Pieske B, Riley JP, Rosano GM, Ruilope LM, Ruschitzka F, Rutten FH, van der Meer P; Authors/Task Force Members; Document Reviewers. 2016 ESC Guidelines for the diagnosis and treatment of acute and chronic heart failure: The Task Force for the diagnosis and treatment of acute and chronic heart failure of the European Society of Cardiology (ESC). Developed with the special contribution of the Heart Failure Association (HFA) of the ESC. Eur J Heart Fail. 2016 Aug;18(8):891-975. doi: 10.1002/ejhf.592. Epub 2016 May 20. No abstract available. PMID 27207191
- [Background] Friedewald VE Jr, Burnett JC Jr, Januzzi JL Jr, Roberts WC, Yancy CW. The editor's roundtable: B-type natriuretic peptide. Am J Cardiol. 2008 Jun 15;101(12):1733-40. doi: 10.1016/j.amjcard.2008.03.017. Epub 2008 Apr 22. No abstract available. PMID 18549849
- [Background] Mueller T, Gegenhuber A, Poelz W, Haltmayer M. Diagnostic accuracy of B type natriuretic peptide and amino terminal proBNP in the emergency diagnosis of heart failure. Heart. 2005 May;91(5):606-12. doi: 10.1136/hrt.2004.037762. PMID 15831643